CLINICAL TRIAL: NCT04854226
Title: Protein Turnover in Preterm Infants - Feeding of Target Fortified Breast Milk With Different Carbohydrate and Fat Composition to Improve Growth
Brief Title: Protein Turnover in Preterm Infants - Feeding of Target Fortified Breast Milk With Different Macronutrient Composition to Improve Growth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paracelsus Medical University (Other)
Collaborators: University Medical Center Rostock (Other); Klinikum Südstadt, Rostock, Germany (Unknown)
Responsible Party: Principal Investigator, Niels Rochow, MD, PhD, Principal Investigator, Paracelsus Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SZ_D_069_20-IX-1
Record Dates: First submitted 2021-04-12; First posted 2021-04-22 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Infant Development; Protein-energy; Imbalance; Protein Deposition
Keywords: protein turnover; growth; tracer; macronutrients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Doctors, nurses and parents are blinded to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Macronutrient_CARB (Experimental): High carbs, low fat composition.
  Interventions: Dietary Supplement: Macronutrients_CARB
- Macronutrient_FAT (Active Comparator): Low carbs, high fat composition.
  Interventions: Dietary Supplement: Macronutrient_FAT

INTERVENTIONS:
Dietary Supplement: Macronutrients_CARB — Breast milk 150 to 170 mL/d; Target fortification: 9.0 g/100mL COH, 3.0 g/100mL protein, 4.0 g/100mL fat, 86.4 kcal/100mL
  Arms: Macronutrient_CARB
Dietary Supplement: Macronutrient_FAT — Breast milk 150 to 170 mL/d; Target fortification: 5.5 g/100mL COH, 3.0 g/100mL protein, 5.5 g/100mL fat, 86 kcal/100mL
  Arms: Macronutrient_FAT

SUMMARY:
The purpose of this study is to measure protein turnover rates in preterm infants.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all parents giving written informed consent the principal investigator will determine the eligibility for study entry. Patients who met the eligibility requirements will be randomized in a double-blind manner in a 1:1 ratio to fortified breast milk with higher fat composition to fortified breast milk with higher carbohydrate composition. Both groups will receive a stable protein composition. The participants will receive the intervention for 3 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 32 weeks
* Enteral nutrition >150 mL / kg / d

Exclusion Criteria:

* gastrointestinal malformations
* Enterostoma
* short bowel syndrome
* necrotizing enterocolitis
* kidney disease
* Foreseeable transfer

Ages: 23 Weeks to 32 Weeks | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
weight gain | daily for 3 weeks
  weight gain in gram
Protein turnover and net protein gain | weekly for 3 weeks
  Tracer N15 labelled amino acids
Protein excretion | weekly for 3 weeks
  Urinary urea in mg/dL and urine volume in mL will be combined to report protein excretion per urine sample (g/kg/d).

SECONDARY OUTCOMES:
Nutritional intake | daily for 3 weeks
  Volume of Breast Milk in mL/kg/d, Lactose in g/100mL, protein g/100mL, fat g/100mL will be combinded to report energy in kcal/kg/d
head circumference | daily for 3 weeks
  in cm
body length | daily for 3 weeks
  in cm
body composition | weekly for 3 weeks
  Fat mass in g, fat-free mass g, volume in L will be combined to report body density in kg/L

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Klinik für Neugeborene, Kinder und Jugendliche Universitätsklinik der Paracelsus Medizinischen Privatuniversität, Nuremberg
  - Universitätsmedizin Rostock Kinder und Jugendklinik, Rostock
  - Klinikum Südstadt Rostock Abteilung für Neonatologie und Neonatologische Intensivmedizin, Rostock

IPD SHARING:
Plan to Share IPD: No